CLINICAL TRIAL: NCT05955872
Title: A Phase 1, Open Label, Randomized, Crossover Study Evaluating the Relative Bioavailability and Food Effect of a VX-147 Test Tablet Formulation Compared to a Reference Tablet Formulation in Healthy Adult Subjects
Brief Title: A Study Evaluating the Relative Bioavailability and Food Effect of a Tablet Formulation of VX-147
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX22-147-010
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Focal Segmental Glomerulosclerosis (FSGS)
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence A: VX-147 (Experimental): Participants will receive VX-147 reference tablet under fasted condition in Treatment Period 1, then VX-147 test tablet under fed condition in Treatment Period 2, and VX-147 test tablet under fasted condition in Treatment Period 3. A washout period of 5 days will be maintained between 3 treatment periods.
  Interventions: Drug: VX-147
- Sequence B: VX-147 (Experimental): Participants will receive VX-147 test tablet under fed condition in Treatment Period 1, then VX-147 test tablet under fasted condition in Treatment Period 2, and VX-147 reference tablet under fasted condition in Treatment Period 3. A washout period of 5 days will be maintained between 3 treatment periods.
  Interventions: Drug: VX-147
- Sequence C: VX-147 (Experimental): Participants will receive VX-147 test tablet under fasted condition in Treatment Period 1, then VX-147 reference tablet under fasted condition in Treatment Period 2, and VX-147 test tablet under fed condition in Treatment Period 3. A washout period of 5 days will be maintained between 3 treatment periods.
  Interventions: Drug: VX-147

INTERVENTIONS:
Drug: VX-147 — Tablets for oral administration.

SUMMARY:
The purpose of the study is to evaluate the relative bioavailability (BA) and the effect of food on the pharmacokinetics (PK), and the safety and tolerability of VX-147 test tablet formulation.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per square meter (kg/m^2), inclusive
* A total body weight greater than 50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-147 Test Compared to VX-147 Reference | From Day 1 up to Day 16
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-147 Test Compared to VX-147 Reference | From Day 1 up to Day 16
Cmax of VX-147 Test Compared Under Fed Versus Fasted State | From Day 1 up to Day 16
AUC(0-inf) of VX-147 Test Compared Under Fed Versus Fasted State | From Day 1 up to Day 16

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious AEs | From Day -1 up to Day 27

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing.